CLINICAL TRIAL: NCT05766956
Title: Effect of Advanced Care at Home vs. Traditional Brick-and-Mortar Hospital Care in Acutely Ill Adults: A Pragmatic Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael J. Maniaci, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-013387
Record Dates: First submitted 2023-03-02; First posted 2023-03-13 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Acute Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Advanced Care at Home (ACH) (Experimental): Patients will receive inpatient hospitalization at home.
  Interventions: Other: Advanced Care at Home (ACH)
- Traditional Inpatient (Brick-and-Mortar) Hospital Care (Active Comparator): Patients will receive inpatient hospitalization at the hospital.
  Interventions: Other: Traditional Brick-and-Mortar Hospitalization

INTERVENTIONS:
Other: Advanced Care at Home (ACH) — Inpatient hospitalization offered in the home setting.
  Arms: Advanced Care at Home (ACH)
Other: Traditional Brick-and-Mortar Hospitalization — Inpatient hospitalization offered in the hospital setting.
  Arms: Traditional Inpatient (Brick-and-Mortar) Hospital Care

SUMMARY:
The purpose of this study is to compare two care delivery models that are currently being implemented in routine practice settings. The findings from this study will inform future clinical decision making, such as which patients might be more suited for which care delivery model.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years of age and older
* Present to one of the participating hospitals
* Have a chief complaint of one of the target diagnoses
* Are within a certain geographical area (based on zip codes)
* Have a health insurance plan that covers ACH services
* Have the capacity to consent or could assent with the consent of a health care proxy who is physically present

Exclusion Criteria:

* Not suitable for ACH or inpatient hospital care as determined by the patient's clinical team
* Do not have the capacity to consent or assent with the assistance of a health care proxy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome is a composite outcome of all-cause mortality | 30 days post-discharge
  The rate of death
30-day readmission | 30 days post-discharge
  Readmission between discharge from ACH/traditional inpatient hospital care and 30 days post-discharge

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Mayo Clinic Health System, Eau Claire, Wisconsin

IPD SHARING:
Plan to Share IPD: No